CLINICAL TRIAL: NCT00005025
Title: A Phase II Trial of In Vivo Gene Therapy With the Herpes Simplex Thymidine Kinase for the Treatment of Ovarian Cancer
Brief Title: Gene Therapy in Treating Women With Refractory or Relapsed Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: John Stoddard Cancer Center at Iowa Methodist Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067546; HGTRI-0105; NCI-V00-1584
Record Dates: First submitted 2000-04-06; First posted 2003-05-05 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2003-03

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Ganciclovir

INTERVENTIONS:
Biological: herpes simplex thymidine kinase
Drug: ganciclovir

SUMMARY:
RATIONALE: Gene therapy may make the body build an immune response to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gene therapy in treating women who have refractory or relapsed ovarian epithelial cancer, fallopian tube cancer, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and safety of in vivo gene therapy with herpes simplex thymidine kinase (HSVtk) vector producer cells (VPC) followed by ganciclovir in women with refractory or relapsed ovarian epithelial adenocarcinoma, fallopian tube cancer, or peritoneal cancer.
* Determine any development of systemic immunity to this regimen or tumor in these patients.
* Determine the toxic effects of intraperitoneal HSVtk VPC in these patients.

OUTLINE: All patients receive an intraperitoneal catheter prior to infusion.

Patients receive herpes simplex thymidine kinase (HSVtk) vector producer cells (VPC) IP over 15-60 minutes on day 0, followed by ganciclovir IV 2 times daily on days 28-41. Treatment repeats for up to 3 courses in patients with stable or responsive disease.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 14-20 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed, refractory or relapsed, ovarian epithelial adenocarcinoma, fallopian tube cancer, or extraovarian peritoneal cancer for which no curative therapy exists

  * Must have tissue available from tumor biopsy to grow tumor cells ex vivo
  * Must have failed standard therapy with both a platinum agent (cisplatin or carboplatin) and paclitaxel
* Site of disease must be less than 5 cm in greatest diameter
* Evaluable disease by CT scan, physical exam, or laparoscopy
* No significant peritoneal fibrosis either from disease or prior surgery

  * Surgical lysis of adhesions allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 2,000/mm3
* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 50,000/mm3
* Hemoglobin at least 8.5 g/dL (without transfusion)

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT or SGPT no greater than 4 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 4 times ULN
* Hepatitis B surface antigen test required prior to study if transaminases greater than 2.0 times ULN
* No hepatitis B surface antigen
* Amylase normal
* PT and PTT normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No cardiac dysfunction by history and exam
* No ischemic heart disease that may be considered anesthetic or operative risk

Pulmonary:

* No lung disease that may be considered anesthetic or operative risk

Other:

* HIV negative
* Not pregnant or nursing
* No acute viral, bacterial, or fungal infection requiring medication within 14 days prior to study
* No patient with greater than 2 L of ascites at the time of intraperitoneal infusion
* No underlying condition that would preclude compliance
* No allergies to study reagent

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No concurrent high dose vitamin regimens

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Charles Joseph Link, MD, Study Chair — John Stoddard Cancer Center at Iowa Methodist Medical Center
Locations (1):
- Human Gene Therapy Research Institute, Des Moines, Iowa, United States